CLINICAL TRIAL: NCT04737759
Title: Taking Care of Us: A Dyadic Intervention for Heart Failure
Brief Title: Taking Care of Us: A Dyadic Intervention for Heart Failure Couples
Acronym: TCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston College (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Karen Lyons, Associate Professor, Boston College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21.074; R21AG068715 (NIH)
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure
Keywords: Couples; Spouses; Dyads
MeSH Terms: conditions — Heart Failure | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taking Care of Us (Experimental): Taking Care of Us involves seven sessions delivered via Zoom to couples over approximately two months. Sessions last approximately 45-60 minutes and are delivered by a trained interventionist. The program is a communication-based, relationship-focused intervention that is strengths-based and fosters new skills to support couples managing heart failure. The goals of the program are to 1) target the couple with heart failure as a team; 2) increase shared appraisal within the couple; 3) improve communication skills within the couple; 4) improve collaboration within the couple and dyadic management of heart failure; 5) improve confidence within the couple; and 6) improve both individual and dyadic health and well-being.
  Interventions: Behavioral: Taking Care of Us
- SUPPORT (Active Comparator): The SUPPORT program involves three sessions delivered via Zoom to couples over approximately two months. Sessions last approximately 45-60 minutes and are delivered by a trained interventionist. This arm is an educational intervention to support management of heart failure.
  Interventions: Other: SUPPORT

INTERVENTIONS:
Behavioral: Taking Care of Us — A social-behavioral intervention that is targeted at the couple living with heart failure and delivered via Zoom.
  Arms: Taking Care of Us
Other: SUPPORT — SUPPORT is an educational counseling intervention that is targeted at the couple living with heart failure and delivered by Zoom.
  Arms: SUPPORT

SUMMARY:
This research study is evaluating the efficacy and feasibility of a novel, dyadic intervention for heart failure couples versus an educational counseling intervention.

DETAILED DESCRIPTION:
There is a critical need for theoretically- and empirically-driven dyadic interventions to improve the outcomes of both adults with heart failure and their partners. The proposed study will evaluate a novel, dyadic program, Taking Care of Us, versus an educational counseling condition using a randomized controlled trial on 72 couples living with heart failure. Both programs are offered via Zoom by trained interventionists and last approximately two months.

Specifically, we will 1) determine the efficacy of the Taking Care of Us intervention on dyadic health; 2) determine the efficacy of the Taking Care of Us intervention on dyadic appraisal and dyadic management; and 3) determine the feasibility and acceptability of the Taking Care of Us intervention.

ELIGIBILITY:
Inclusion Criteria: Adults with Heart Failure:

* Diagnosis of heart failure for at least three months
* Current heart failure symptoms (i.e., NYHA Class II-III; AHA/ACC Stage C)
* Age greater than or equal to 18 years
* Willing and able to provide informed consent
* Reachable by telephone/email
* Access to device with camera (e.g., computer, tablet) to participate in Zoom sessions
* Have a co-residing spouse/unmarried partner willing to participate

Inclusion Criteria: Spouses/Partners:

* Age greater than or equal to 18 years
* Co-residing with the adult with heart failure at time of recruitment
* Have lived with the adult with heart failure for at least one year
* Willing and able to provide informed consent

Exclusion Criteria:

* Major and uncorrected hearing impairment
* Significant cognitive impairment
* Heart transplantation/mechanical circulatory support prior to enrollment
* Concomitant terminal illness that would impede participation
* Active psychosis or severe substance abuse that would impair the ability to complete the study
* Inability to complete the requirements of the study, including enrolment in an additional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen S Lyons, PhD, Principal Investigator — Boston College; Christopher S Lee, PhD, RN, Principal Investigator — Boston College
Locations (2):
- United States (2):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston College, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lyons KS, Whitlatch CJ, Vest AR, Upshaw JN, Hutton Johnson S, Walters A, Lee CS. Feasibility, Acceptability, and Preliminary Efficacy of the Taking Care of Us Intervention for Couples Living With Heart Failure. Innov Aging. 2024 Dec 7;9(1):igae106. doi: 10.1093/geroni/igae106. eCollection 2025. PMID 39790834
- [Derived] Lyons KS, Whitlatch CJ, Vest AR, Upshaw JN, Johnson SH, Morelock J, Lee CS. Taking Care of Us(c) (TCU) study protocol: feasibility and acceptability of a dyadic intervention for couples living with heart failure. Pilot Feasibility Stud. 2023 Jan 25;9(1):16. doi: 10.1186/s40814-023-01249-7. PMID 36698174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 74 participants (37 couples). Recruitment began February 2021. Participants completed consent and enrolled between July 2021 and November 2022. Study investigators at Tufts Medical Center Heart Failure clinic, Boston, MA provided patients with recruitment materials in-person (when possible) and via mailings. Recruitment also involved community outreach locally (e.g., councils on aging, newsletters, media), nationally via social media, websites and clinical colleagues.
Period: Overall Study
Arm/Group | Taking Care of Us | SUPPORT
Started | 36 | 38
Adults With Heart Failure | 18 | 19
Spouse/Partners | 18 | 19
Completed | 16 (16 paticipants (8 adults with heart failure and 8 partners)) | 22 (22 participants (11 adults with heart failure and 11 partners))
Not Completed | 20 | 16
Not completed — Patient and spouse withdrew as adult with heart failure too sick/health decline | 12 | 4
Not completed — Death | 2 | 0
Not completed — spouse dropped when adult with heart failure died | 2 | 0
Not completed — Lost to Follow-up | 4 | 12

BASELINE CHARACTERISTICS:
Population: 18 couples consisting of 18 adults with heart failure and 18 spouse/partners for a total of 36 participants in Taking Care of Us 19 couples consisting of 19 adults with heart failure and 19 spouse/partners for a total of 38 participants in SUPPORT
Groups:
- Total: Total of all reporting groups
Arm/Group | Taking Care of Us | SUPPORT | Total
Number analyzed (Participants) | 36 | 38 | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: We had 37 couples participate (37 adults with heart failure and 37 spouse/partners)
  Years
    Patient with heart failure age: number analyzed (Participants) | 18 | 19 | 37
    Patient with heart failure age | 64.61 (15.15) | 68.03 (12.33) | 66.32 (13.72)
    Spouse/partner age: number analyzed (Participants) | 18 | 19 | 37
    Spouse/partner age | 61.67 (15.03) | 64.26 (10.35) | 63.00 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 37 couples for total of 74 participants (37 patients and 37 partners)
  Participants
    Patient with heart failure: number analyzed (Participants) | 18 | 19 | 37
    Patient with heart failure: Female | 4 | 4 | 8
    Patient with heart failure: Male | 14 | 15 | 29
    Spouse/Partner: number analyzed (Participants) | 18 | 19 | 37
    Spouse/Partner: Female | 14 | 15 | 29
    Spouse/Partner: Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 37 couples
  Participants
    Patient with heart failure: number analyzed (Participants) | 18 | 19 | 37
    Patient with heart failure: Hispanic or Latino | 0 | 1 | 1
    Patient with heart failure: Not Hispanic or Latino | 18 | 18 | 36
    Patient with heart failure: Unknown or Not Reported | 0 | 0 | 0
    Spouse/Partner: number analyzed (Participants) | 18 | 19 | 37
    Spouse/Partner: Hispanic or Latino | 1 | 0 | 1
    Spouse/Partner: Not Hispanic or Latino | 17 | 19 | 36
    Spouse/Partner: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 37 couples (37 patients and 37 partners)
  Participants
    Patient with heart failure: number analyzed (Participants) | 18 | 19 | 37
    Patient with heart failure: American Indian or Alaska Native | 0 | 0 | 0
    Patient with heart failure: Asian | 0 | 0 | 0
    Patient with heart failure: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Patient with heart failure: Black or African American | 0 | 0 | 0
    Patient with heart failure: White | 17 | 18 | 35
    Patient with heart failure: More than one race | 1 | 1 | 2
    Patient with heart failure: Unknown or Not Reported | 0 | 0 | 0
    Spouse/partner: number analyzed (Participants) | 18 | 19 | 37
    Spouse/partner: American Indian or Alaska Native | 0 | 0 | 0
    Spouse/partner: Asian | 0 | 0 | 0
    Spouse/partner: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Spouse/partner: Black or African American | 0 | 0 | 0
    Spouse/partner: White | 18 | 19 | 37
    Spouse/partner: More than one race | 0 | 0 | 0
    Spouse/partner: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 38 | 74
Education Level [Count of Participants; unit: Participants] — Number who attended some college Population: 37 couples (37 patients and 37 partners)
  Participants
    Patients with heart failure: number analyzed (Participants) | 18 | 19 | 37
    Patients with heart failure | 11 | 16 | 27
    Spouse/Partners: number analyzed (Participants) | 18 | 19 | 37
    Spouse/Partners | 14 | 16 | 30
Heart failure severity [Mean (Standard Deviation); unit: units on a scale] — Self-reported 1 (can do ordinary physical activities without symptoms); 2 (ordinary physical activities causes symptoms); 3 (less than ordinary physical activity causes symptoms); 4 (experience symptoms at rest). Population: Only patients self-reported on heart failure severity.
  units on a scale
    number analyzed (Participants) | 18 | 19 | 37
    (all) | 2.28 (0.9) | 2.21 (0.86) | 2.24 (0.86)
Financial insecurity [Count of Participants; unit: Participants] — Measure of financial security: 1 (more than enough to make ends meet); 2 (enough to make ends meet); 3 (not enough to make ends meet). Percentage reporting a value of "3" Population: Self-reported by patients
  Participants
    number analyzed (Participants) | 18 | 19 | 37
    (all) | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Quality of Life Scores in Couples in the TCU vs SUPPORT Condition.
Description: Physical quality of life score from the 10-item PROMIS Global Health Short Form. 4 items recoded to 1-5 scale for potential range of 1-20. Higher scores indicate better physical quality of life.
Time Frame: 5 months after baseline
Population: Intent to treat: All participants who were assigned to an arm included. Last observation point carried forward (LOCF) imputation method used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | 1.28 (1.74) | -0.03 (1.51)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | 0.59 (1.42) | -0.63 (1.92)

2. Primary Outcome: Change in Mental Quality of Life Scores in Couples in the TCU vs SUPPORT Condition.
Description: Mental quality of life score from the 10-item PROMIS Global Health Short Form. 4 items recoded to 1-5 scale for potential range of 1-20. Higher scores indicate better mental quality of life.
Time Frame: 5 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | 0.39 (1.58) | 0.34 (1.83)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | 0.50 (1.58) | -0.21 (1.84)

3. Secondary Outcome: Change in Depressive Symptom Scores in Couples in the TCU vs SUPPORT Condition.
Description: Center for Epidemiological Studies Depression CESD 20-item measure. Items are on a 0-3 scale with potential range of 0-60 with higher scores indicating more depressive symptoms.
Time Frame: 5 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | -5.83 (11.17) | -0.74 (2.71)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | -0.44 (3.78) | -0.40 (3.64)

4. Secondary Outcome: Change in Care Strain Scores in Spouses in the TCU vs SUPPORT Condition.
Description: The 16-item Multidimensional Caregiver Strain Index measures physical, social, interpersonal strain and time constraints and demands related to providing care on a 1-5 scale. Potential range of scores is 16-80 with higher scores indicating greater strain.
Time Frame: 5 months after baseline
Population: Intent to treat: All spouse/partners (18 in Taking Care of Us and 19 in SUPPORT) who were assigned to an arm included. Last observation point carried forward (LOCF) imputation method used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 18 | 19
units on a scale | -1.72 (5.98) | 1.32 (5.57)

5. Secondary Outcome: Change in Heart Failure Related Quality of Life Scores in Persons With Heart Failure in the TCU vs SUPPORT Condition
Description: Total quality of life score assessed by the 12-item Kansas City Cardiomyopathy Questionnaire. Items are converted to a 0-100 scale with higher scores indicating better heart failure related quality of life.
Time Frame: 5 months after baseline
Population: Intent to treat: All participants who were assigned to an arm included. Last observation point carried forward (LOCF) imputation method used. Measure only completed by the 37 patients with heart failure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 18 | 19
units on a scale | 5.90 (13.23) | -0.82 (15.72)

6. Secondary Outcome: Change in Difference in Dyspnea Scores in the TCU vs SUPPORT Condition
Description: Patient dyspnea scores assessed by the 6-item Heart Failure Somatic Perception Scale. Items ask about how much the person was bothered by dyspnea during the last week on a 0 (not at all) to 5 (extremely bothersome) scale for a potential range of 0-30. Higher scores indicate greater dyspnea. It was not possible to examine changes in incongruence within couples due to small sample so between-group differences with patients and spouses (reporting their perception of patient's dyspnea) were calculated.
Time Frame: 5 months after baseline
Population: Intent to treat: All participants who were assigned to an arm included. Last observation point carried forward (LOCF) imputation method used. Only patients with heart failure self-reported dyspnea; partners reported their perception of the patient's dyspnea.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | -2.06 (5.39) | 0.11 (4.56)
  Report of spouse/partner: number analyzed (Participants) | 18 | 19
  Report of spouse/partner | -1.83 (3.81) | 0.47 (5.78)

7. Secondary Outcome: Change in Difference in Pain Interference Scores in Couples in the TCU vs SUPPORT Condition
Description: Pain interference was assessed using the six-item PROMIS pain interference scale with items ranging from 1-5 for a potential range of 6-30. Higher scores indicate more pain interference. It was not possible to examine changes in incongruence within couples due to small sample so between-group differences with patients and spouses (reporting their perception of patient's pain interference) were calculated.
Time Frame: 5 months after baseline
Population: Intent to treat: All participants who were assigned to an arm included. Last observation point carried forward (LOCF) imputation method used. Only patients with heart failure self-reported pain interference; partners reported their perception of the patient's pain interference.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | -3.50 (4.32) | 1.68 (4.28)
  Report of spouse/partner: number analyzed (Participants) | 18 | 19
  Report of spouse/partner | -1.61 (5.45) | 2.47 (8.61)

8. Secondary Outcome: Change in Difference in Fatigue Scores in Couples in the TCU vs SUPPORT Condition.
Description: Fatigue was assessed using the eight-item PROMIS fatigue scale with items on a 1-5 scale for a potential range of 8-40. Higher scored indicate more fatigue. It was not possible to examine changes in incongruence within couples due to small sample so between-group differences with patients and spouses (reporting their perception of patient's fatigue) were calculated.
Time Frame: 5 months baseline
Population: It was not possible to examine changes in incongruence within couples due to small sample so between-group differences with patients and spouses (reporting their perception of patient's fatigue) were calculated. Intent to treat: All participants who were assigned to an arm included. Last observation point carried forward (LOCF) imputation method used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | -2.33 (5.65) | -0.21 (6.76)
  Report of spouse/partner: number analyzed (Participants) | 18 | 19
  Report of spouse/partner | -3.06 (5.52) | -0.42 (6.14)

9. Secondary Outcome: Change in Collaboration Scores in Couples in the TCU vs SUPPORT Condition
Description: Collaborative symptom management was assessed using the six-item Stanford Chronic Disease Self-Management measure with items reworded to ask how much couples worked together to prevent symptoms (e.g., fatigue, pain, emotional distress) from interfering with what the person with heart failure wanted to do or to reduce the need to see a provider on a 1 (never) to 10 (always) scale. Average summary scores had the potential to range from 1-10 with higher scores indicating greater collaborative management.
Time Frame: 5 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | 1.13 (2.33) | 0.40 (2.29)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | 1.20 (1.65) | 0.28 (1.84)

10. Secondary Outcome: Change in Confidence Scores in Couples in the TCU vs SUPPORT Condition
Description: Confidence was measured using the 6-item Stanford Chronic Disease Self-Management measure to assess confidence to manage six aspects of the illness (e.g., fatigue, emotional distress) on a 1 (no confidence) to 10 (a great deal of confidence) scale. Summary scores were calculated by average the six items for a potential range of 1-10.Higher scores indicate greater confidence.
Time Frame: 5 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | 0.33 (1.48) | -0.06 (1.96)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | 0.51 (1.52) | -0.23 (2.39)

11. Secondary Outcome: Change in Communication Scores on the Active Engagement Subscale in Couples in the TCU vs SUPPORT Condition
Description: Communication within the couple was assessed using both scales from the Dyadic Coping measure. Active engagement has five items that ask about how much one's partner engages in open communication and support on a 1-5 scale for a possible range of 5-25. Higher scores indicate one's partner has a higher level of active engagement.
Time Frame: 5 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | 1.11 (2.72) | -0.58 (3.20)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | 2.17 (3.79) | 0.74 (1.91)

12. Secondary Outcome: Change in Communication Scores on the Protective Buffering Subscale in Couples in the TCU vs SUPPORT Condition
Description: Communication within the couple was assessed using both scales from the Dyadic Coping measure. Protective buffering has six items that ask about how much one's partner engages in hiding concerns and denying worries on a 1-5 scale for a possible range of 6-30. Higher scores indicate one's partner has a higher level of protective buffering.
Time Frame: 5 months after baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us | SUPPORT
Number analyzed (Participants) | 36 | 38
units on a scale
  Patients with heart failure: number analyzed (Participants) | 18 | 19
  Patients with heart failure | -1.39 (2.93) | 0.05 (2.12)
  Spouse/partner: number analyzed (Participants) | 18 | 19
  Spouse/partner | 0.00 (4.55) | 0.42 (2.22)

13. Other Pre Specified Outcome: Satisfaction Scores in Couples in the TCU Condition as a Measure of Acceptability.
Description: Satisfaction with the assigned program was assessed with a Likert item adapted from other intervention work about the benefits and drawbacks of the program. Participants were asked to rate their satisfaction with the overall program on a 1 to 4 scale with higher scores indicating greater satisfaction.
Time Frame: 5 months after baseline
Population: Data from all those in the Taking Care of Us arm, who complete the 5 month follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taking Care of Us
Number analyzed (Participants) | 16
units on a scale
  Patients with heart failure: number analyzed (Participants) | 8
  Patients with heart failure | 3.63 (1.01)
  Spouse/partners: number analyzed (Participants) | 8
  Spouse/partners | 3.57 (0.79)

ADVERSE EVENTS:
Time Frame: 5 months (from enrollment until 5 month follow-up.
Arm/Group | Taking Care of Us | SUPPORT
All-Cause Mortality (participants affected / at risk) | 2/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/59/NCT04737759/Prot_SAP_000.pdf